CLINICAL TRIAL: NCT03527810
Title: Hiatal Interrogation in Sleeve Gastrectomy (HIATUS):a Clinical Trial
Brief Title: Hiatal Interrogation in Sleeve Gastrectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interim analysis of the data was not supportive of continuing the study.
Sponsor: Miguel Burch (Other)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor-Investigator, Miguel Burch, Associate Director, Minimally Invasive Surgery, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro47769
Record Dates: First submitted 2018-03-22; First posted 2018-05-17 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Sleeve Gastrectomy
Keywords: sleeve gastrectomy; hiatal interrogation; GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeve Gastrectomy With Interrogation of Hiatus (Experimental): In those randomized to interrogation, the hiatus will be opened posteriorly during surgical procedure intervention with preservation of the phreno-esophageal ligament where possible, as per standard described techniques. Dissection into the mediastinum will be stopped if no hernia is seen or when appropriate intra-abdominal length of 2 cm of esophagus is created. Once opened, the Hiatal Surface Area will be measured, calculated and recorded and when possible, a photo taken of the area. Repair of the crura will then be performed around the sizing tube used to create the sleeve with enough space to allow a 5 mm instrument to be easily inserted. Permanent sutures will be placed posterior to the esophagus.
  Interventions: Procedure: Sleeve Gastrectomy With Interrogation of Hiatus
- Sleeve Gastrectomy Without Interrogation of Hiatus (Active Comparator): In those randomized without interrogation, the stomach is reduced to about 15% of its original size, by surgical removal of a large portion of the stomach along the greater curvature. The procedure involves a longitudinal resection of the stomach starting from the antrum at the point 5-6 cm from the pylorus and finishing at the fundus close to the cardia.[1] The remaining gastric sleeve is calibrated with a bougie. Most surgeons prefer to use a bougie between 36-40 Fr with the procedure and the ideal approximate remaining size of the stomach after the procedure is about 150 mL.
  Interventions: Procedure: Sleeve Gastrectomy Without Interrogation of Hiatus

INTERVENTIONS:
Procedure: Sleeve Gastrectomy Without Interrogation of Hiatus — Weight-loss procedure to reduce the stomach.
  Arms: Sleeve Gastrectomy Without Interrogation of Hiatus
Procedure: Sleeve Gastrectomy With Interrogation of Hiatus — Weight-loss procedure to reduce the stomach with hiatal repair.
  Arms: Sleeve Gastrectomy With Interrogation of Hiatus

SUMMARY:
The subject will undergo standard pre-operative preparation. Subjects will be evaluated for the presence of bothersome GERD symptoms by GERD questionnaires and use of Proton-Pump Inhibitor (PPI) medications. Those eligible will be approached at their preoperative appointment about participation in the study and consent will be reviewed with subject. Signed consent will be collected from the subject prior to entry into the operating room. After induction of anesthesia, the subject will be randomized to sleeve gastrectomy with or without interrogation of the hiatus.

The SG will be performed as per standard approaches already described. In those randomized to interrogation, the hiatus will be opened posteriorly with preservation of the phreno-esophageal ligament where possible, as per standard described techniques. Dissection into the mediastinum will be stopped if no hernia is seen or when appropriate intra-abdominal length of 2 cm of esophagus is created. Once opened, the Hiatal Surface Area (appendix B)17 will be measured, calculated and recorded and when possible, a photo taken of the area. Repair of the crura will then be performed around the sizing tube used to create the sleeve with enough space to allow a 5 mm instrument to be easily inserted. Permanent sutures will be placed posterior to the esophagus.

Subjects will be recovered and be discharged per standard protocol. Evaluation for reflux will be conducted pre-operatively and then 3, 6, 12 and 24 months (+/- 30 days) after surgery or on demand if symptoms occur between follow up periods. Many groups advocate the use of PPI for the first 30 days after bariatric surgery - accordingly assessments of reflux will not occur until 3 months post operatively when most groups stop prophylactic PPI use. A visit within the first 30 days after surgery (+/- 15 days) should occur to evaluate for potential complications of surgery.

DETAILED DESCRIPTION:
The obesity epidemic continues to exist as nearly one third of the adult population in the United States is reported to be obese1. Bariatric surgery remains the most effective method of achieving long-term weight loss among obese individuals. The remarkable success of weight loss surgery in ameliorating obesity and its related comorbid conditions has been tempered by procedure specific side-effect profiles. Gastro-esophageal reflux disease (GERD), a condition which develops when the reflux of stomach contents causes troublesome heartburn or regurgitation symptoms greater than twice a week is a known complication of bariatric surgery and remains a controversial topic among bariatric surgeons.2 The prevalence of GERD in the general Western population is between 10 and 20% 3, whereas the incidence of reflux among the obese population has been reported to be as high as 61%. 4

The safety and maintenance of native intestinal anatomy by the sleeve gastrectomy (SG) has recently made this surgery the most popular operation for weight loss in America 5. The operation, which was originally described as the first stage of a biliopancreatic diversion - duodenal switch, consists of removing approximately 60% of the native stomach. Specifically, the bulbous greater curvature and a portion of the antrum is removed, leaving behind a long, thin banana shaped reservoir with a capacity between 100 and 150 mL. 6 This new stomach offers excellent weight loss and also minimal anatomic rearrangement when compared to the traditional gastric bypass.

Although some authors have reported an improvement in GERD symptoms after SG many studies have demonstrated an increase in GERD symptoms9-14. Particularly concerning is the development of de-novo GERD symptoms after surgery, which has recently been reported to occur in up to 36% of patients when measured objectively.15 In some, GERD symptoms are severe enough, despite medication, that corrective operations are required. The need for further re-operative surgery carries along with it the risk for additional perioperative morbidity from gastrointestinal leaks or bleeding as well as further time off work and rehabilitation.

Various mechanisms have been proposed to explain the development of GERD after SG. Some authors postulate that the new shape of the stomach, increased intra-gastric pressure, decrease in the lower esophageal sphincter resting pressure or development of a hiatal hernia may lead to new or worsening GERD. The International Sleeve Gastrectomy Expert Panel recommend aggressively inspecting for and repairing an occult hiatal hernia to decrease the incidence of post-operative GERD.17 This call for "aggressive inspection" has led many surgeons to open the phrenoesophageal ligament and, in a sense, create a small hernia defect which is then sutured closed more tightly. Some believe aggressive interrogation of the hiatus may lead to disruption of the integrity of the sling fibers of Helvetius at the esophagogastric junction, thus contributing to the incidence of new or worsening post-operative GERD. Still, others propose that the main mechanism of GERD reduction is weight loss and not the re-creation of the extrinsic anti-reflux valve.

Whether one should aggressively interrogate and subsequently repair the hiatus during a SG remains controversial. To our knowledge, there are no randomized studies to demonstrate superiority of either approach. The aim is to compare the rates of GERD (de-novo or worsening) in patients undergoing SG between one group receiving hiatal interrogation and repair and the other not having hiatal interrogation at all. Patient are randomized who either have a small hiatal hernia (<2cm) or do not have a hiatal hernia seen on preoperative testing to either hiatal interrogation with cruroplasty of the hiatus or no interrogation. By the end of the study, the study team will be able to provide a recommendation as to whether patients with no or a small hernia undergoing SG should routinely undergo simultaneous hiatal interrogation and repair with the goal of reducing the incidence of PPI de-novo GERD after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient deemed a candidate for Sleeve Gastrectomy.
2. Age 18 years or older.
3. Body Mass Index equal or greater to 40 without comorbidities OR Body Mass Index equal or greater than 35 with at least one obesity co-morbidity.

Exclusion Criteria:

1. The presence of one or more of the following will be reason for exclusion:

   1. Daily Proton Pump Inhibitor or H2 blocker use for typical GERD symptoms during Screening day to Surgery day
   2. GERD Health Related Quality of Life (HRQL) questionnaire score greater than or equal to 15.
2. Hiatal hernia greater than 2cm by either preoperative endoscopy or Upper gastrointestinal (UGI) within one year of evaluation for bariatric surgery.
3. The Los Angeles classification of the severity of reflux esophagitis: C,D
4. Barrett's esophagus
5. Dysphagia with poor esophageal function measured by motility testing.
6. Does not meet National Institute of Health's weight loss surgery criteria.
7. Inability to commit to no pregnancy for 18 months post operatively.
8. Gastroparesis as defined by 4 hour nuclear emptying study.
9. Previous bariatric surgery.
10. Eosinophilia esophagitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Change in patients dependent on proton pump inhibitors therapy for confirmed GERD. | 6 months
  Statistically significant change in total patients on PPI therapy for confirmed GERD (by either questionnaire or pH test confirmed GERD).

SECONDARY OUTCOMES:
Time free from GERD symptoms compared between both groups | 24 months
  number of months
Time free from GERD medications compared between both groups | 24 months
  number of months
Number of patients with symptomatic hiatal hernias at 24 months | 24 months
  number of patients
Number of patients requiring secondary procedures for reflux at 12, 24 months | 12, 24 months
  number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Burch, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No